CLINICAL TRIAL: NCT00994253
Title: A Prospective, Randomized, Open-label Clinical Trial to Evaluate the Effect of Tekturna (Aliskiren), Angiotensin Inhibitors, Diuretics, and Calcium Channel Blockers on Coronary Flow Reserve in Patients With Type II Diabetes and Hypertension
Brief Title: Evaluating the Effect of Aliskiren Versus HCTZ on Coronary Flow Reserve in Hypertensive Type II Diabetics
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to safety concerns re: the concomitant use of aliskiren with an ACEi or ARB.
Sponsor: Corewell Health East (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Pam Marcovitz, MD, Principal Investigator, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-083
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Hypertension; Diabetes Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Experimental): Aliskiren will be prescribed at 150mg po per day. If the subjects blood pressure is not controlled by week 5 the dose will be increased to 300mg po per day.
  Patients will be assigned to the treatment arm containing aliskiren. The prescribed drugs will include: Lisinopril 40mg + amlo 5mg + aliskiren 150-300mg
  Interventions: Drug: Aliskiren
- Hydrochlorothiazide (Active Comparator): HCTZ will be prescribed at 12.5 po per day. If the subjects blood pressure is not controlled by week 5 the dose will be increased to 25mg po per day.
  Patients will be assigned to the treatment arm containing HCTZ. The prescribed drugs will include: Lisinopril 40mg + amlo 5mg + HCTZ 12.5-25mg
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Aliskiren — Aliskiren will be prescribed at 150mg po per day. If the subjects blood pressure is not controlled by week 5 the dose will be increased to 300mg po per day. All subjects will be prescribed lisinopril 40mg and amlodipine 5mg po daily.
  Other Names: Tekturna
  Arms: Aliskiren
Drug: Hydrochlorothiazide — Hydrochlorothiazide will be prescribed at 12.5 po per day. If the subjects blood pressure is not controlled by week 5 the dose will be increased to 25mg po per day. All subjects will be prescribed lisinopril 40mg and amlodipine 5mg po daily
  Other Names: HCTZ
  Arms: Hydrochlorothiazide

SUMMARY:
The purpose of this study is to assess the effect of Tekturna (aliskiren), in combination with an ACE and calcium channel blocker in hypertensive patients diagnosed with Type II diabetes.

DETAILED DESCRIPTION:
This study focuses on diabetic patients who are already on any blood pressure-lowering medication (excluding Tekturna) in addition to either an ACE inhibitor or an ARB (angiotensin receptor blocker) and still have a blood pressure greater than 130/80 mm Hg. The purpose of the study is to compare the effects of two different blood pressure treatment regimens, each containing three medications, on heart function in diabetics with uncontrolled hypertension. The two treatments are 1) lisinopril (an ACE inhibitor that works by reducing blood pressure) plus amlodipine (a calcium channel blocker that reduces blood pressure) plus aliskiren (a renin inhibitor, which also reduces blood pressure), or 2) lisinopril plus amlodipine plus hydrochlorothiazide (a diuretic, or "water pill"). Participants will have their coronary flow reserve - which is a measure of coronary vessel function, a predictor of future cardiovascular events - and a number of cardiovascular biomarkers in blood and urine at baseline and after 6 months of treatment. In this manner hydrochlorothiazide will be compared with aliskiren, which researchers think will have a better effect on heart artery blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Diagnosed with Type II Diabetes and Hypertension
* Taking either ACE or ARB in addition to any other antihypertensive medication excluding aliskiren
* Blood Pressure >130/80

Exclusion Criteria:

* Serum Potassium >5.2 mmol/L
* History of any cardiovascular event (stroke, TIA, unstable angina, CABG, percutaneous coronary intervention, hospitalization due to HF) during the 3 months prior to Visit 1.
* History of MI
* Documented ejection fraction of <50%
* Hypertension (at Screening): any patient with msSBP ≥ 180 mmHg or msDBP ≥ 110 mmHg
* Congestive Heart Failure NYHA class III and IV
* Concomitant treatment with two (2) or more renin-angiotensin-aldosterone system blocking agents, e.g. ACE inhibitor, ARB or aldosterone-antagonist.
* Unstable serum creatinine
* Second (II) or third (III) degree heart block without a pacemaker
* Concurrent potentially life threatening arrythmia or other uncontrolled arrythmia
* Clinically significant valvular heart disease
* Known renal artery stenosis
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of the study drugs including, but not limited to, any of the following:

  * History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection (patients with previous bariatric surgery>6 months prior to Visit 1 are allowed to participate).
  * Any history of pancreatic injury, pancreatitis or evidence of impaired pancreatic function/injury as indicated by abnormal lipase or amylase.
  * Evidence of hepatic disease as determined by any one of the following: SGPT value exceeding 3x Upper Limit of Normal (ULN) at Visit 1, a history of hepatic encephalopathy, a history of cirrhosis, esophageal varices, or a history of portocaval shunt.
* History of malignancy other than basal cell skin cancer that is likely to reduce the subject's life span to less than 2 years.
* Any concurrent life threatening condition with a life expectancy less than 2 years
* History or evidence of drug or alcohol abuse with the last 12 months
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* History of hypersensitively to any of the study drugs or to medications belonging to the same therapeutic class as the study drugs as well as known or suspected contraindications to the study drugs
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* Any condition that in the opinion of the investigator would jeopardized the evaluation of efficacy or safety
* Persons directly involved in the execution of this protocol
* Pregnant or nursing (lactating) women
* Women of Child Bearing Potential unless post menopausal for at least one year, surgically sterile or using effective methods of contraception as defined by local Health Authorities.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08 (Estimated); Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the effect of a multimodal drug therapy regimen including the renin inhibitor Tekturna (aliskiren), an ACE inhibitor, and a calcium channel blocker on coronary flow reserve (CFR) in hypertensive Type II diabetics. | 6 months
  CFR will be assessed by a PET-based imaging technique.

SECONDARY OUTCOMES:
Secondary measures include evaluation of serum and urine biomarkers related to endothelial function, the renin-angiotensin system, oxidative stress, and inflammation. | 6 months
  Biomarkers include asymmetric dimethylarginine, B-type natriuretic peptide, plasma renin activity, high-sensitivity C-reactive protein, adiponectin, aldosterone, angiotensinogen, and hemoglobin A1c.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela A Marcovitz, MD, Principal Investigator — Beaumont Health System, Royal Oak
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No